CLINICAL TRIAL: NCT01115049
Title: Evaluation of the Efficacy of a Hexetidine- and Chlorobutanol-based Mouthwash in the Symptomatic Treatment of Oral Lesions Due to Removable Prostheses: a Prospective, Randomized, Triple-blind Controlled Clinical Trial
Brief Title: Hexetidine and Chlorobutanol for Lesions Due to Prostheses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Fernando Zarone, MD, DDS, Professor and Chair, University "Federico II" of Naples, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FEDII_RS_1
Record Dates: First submitted 2010-04-21; First posted 2010-05-03 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2010-04

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Chlorobutanol; Hexetidine; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental mouthwash (Experimental): The experimental mouthwash (Buccagel®, Curaden Healthcare, Saronno, Italy) was made up of: purified water, dicaprylyl-ether, coco-caprylate caprate, xylitol, glyceryl-stearate, ceteareth-20, ceteareth-12, cetyl-palmitate, cetearyl-alcohol, chlorobutanol, aroma, hexetidine, methylparaben, propylparaben, sodium saccharin, citric acid and colorant C.I. 16255.
  Interventions: Drug: chlorobutanol, hexetidine
- Chlorexidine-based mouthwash (Active Comparator): A conventional commercial mouthwash (Curasept® ADS 0.20%, Curaden Healthcare, Saronno, Italy) made up of: water, xylitol, propylenglycol, Peg-40 of hydrogenated ricin oil, ascorbic acid, chlorhexidine digluconate, aroma, poloxamer 407, sodium metabisulfite, sodium citrate and colorant C.I. 42090.
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: chlorobutanol, hexetidine — 3 times per day (after breakfast, lunch and dinner) for 1 minute with 15 ml of mouthwash
  Other Names: Curasept® ADS 0.20%, Curaden Healthcare
  Arms: Experimental mouthwash
Drug: Chlorhexidine — 3 times per day (after breakfast, lunch and dinner) for 1 minute with 15 ml of mouthwash
  Other Names: Curasept® ADS 0.20%, Curaden Healthcare
  Arms: Chlorexidine-based mouthwash

SUMMARY:
Objectives: The study aimed at assessing the efficacy of a new mouthwash in treating oral lesions due to removable prostheses.

Methods: The present prospective randomized clinical trial was performed on 44 patients. The experimentation lasted for 4 weeks and 4 operators participated. The effects of the mouthwash were evaluated subjectively and objectively, with questionnaires, Visual Analogic Scales and clinical examinations. The results were statistically analyzed. The following variables were recorded: presence of mucosal lesions due to incongruous removable prostheses and lasting of pain after rinsing.

DETAILED DESCRIPTION:
The aim of the present prospective, randomized, triple-blind controlled clinical trial was to evaluate the efficacy of an innovative mouthwash (emulsion) in the treatment of lesions of oral mucosae due to removable prostheses. The tested preparation contained two active molecules: a topical antiseptic (0.1% hexetidine) and a local anesthetic (0.5% chlorobutanol).

ELIGIBILITY:
Inclusion Criteria:

* Use of removable partial or complete dentures;
* Presence of lesions of oral mucosae due to dentures;
* Absence of any concomitant local or systemic pathology;
* Absence of pregnancy or breastfeeding;
* Negative allergic anamnesis;
* Negative anamnesis for recurrent aphthous stomatitis;
* No taking medicines with potential pharmacologic interactions with molecules to be tested;
* No taking antibiotics and/or painkillers for at least 6 months before entering the experimentation;
* Good oral hygiene with a full-mouth plaque score ≤25%;
* Non smoking or light smoking (≤10 cigarettes/day) status.

Exclusion Criteria:

Missing one or more of the above described conditions automatically excluded a subject from the study.

Ages: 37 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of tolerability | Weekly
  Presence of mucosal lesions due to incongruous removable prostheses.

SECONDARY OUTCOMES:
Pain scores on the visual analogue scale | Weekly
  Lasting of painful symptomatology after rinsing.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Zarone, MD, DDS, Study Director — University "Federco II" of Naples, Italy
Locations (1):
- University "Federico II", Department of Prosthodontics, Naples, Italy